CLINICAL TRIAL: NCT06349018
Title: The Effects of Isotonic Beetroot Supplementation on Sprint Interval Exercise Performance.
Brief Title: Effects of Isotonic Beetroot Supplementation on Sprint Interval Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Stephen Burns, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB-2023-972
Record Dates: First submitted 2024-02-20; First posted 2024-04-05 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Exercise Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both isotonic drinks (high nitrate or no nitrate) are deidentified and labelled (coded) by a third party not involved with the research. Randomization and allocation are completed by a third party not involved in the testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High nitrate (Experimental): High nitrate isotonic drink
  Interventions: Other: Dietary Supplement: High nitrate isotonic drink
- No nitrate (Active Comparator): No nitrate isotonic drink
  Interventions: Other: Dietary Supplement: No nitrate isotonic drink

INTERVENTIONS:
Other: Dietary Supplement: High nitrate isotonic drink — High nitrate (12.9 mmol) drink with carbohydrate and minerals
  Arms: High nitrate
Other: Dietary Supplement: No nitrate isotonic drink — Carbohydrate and mineral isotonic drink
  Arms: No nitrate

SUMMARY:
This study aims to examine the effects of dietary nitrate supplementation via beetroot juice on sprint interval cycling exercise performance. Twenty-four participants (male or female) will undertake a randomized, crossover trial where they consume either (i) an isotonic beetroot juice drink containing nitrate (12.9 mmol) for 5 days or (ii) an isotonic sports drink (no nitrate) for 5 days. On Day 5 of each trial, participants will come to the laboratory and 2 hours after consuming their allocated drink will complete a 6 bouts of sprint interval exercise. Power output during cycling will be measured as the primary outcome measure. Salivary and plasma measures of nitrate and nitrite will be taken over the course of the morning on Day 5. After a 5-day washout period participants will crossover and begin their second trial.

DETAILED DESCRIPTION:
This study aims to examine the effects of dietary nitrate supplementation via beetroot juice on sprint interval cycling exercise performance. Twenty-four participants (male or female) will undertake a randomized, crossover trial where they consume either (i) an isotonic beetroot juice drink containing nitrate (12.9 mmol) for 5 days or (ii) an isotonic sports drink (no nitrate) for 5 days. Drinks will be equivalent in isotonicity and colored the same so that participants and investigators will be blinded to each trial. Randomization and drink allocation will be completed by a third person not associated with the study team. On Day 5 of each trial, participants will come to the laboratory and 2 hours after consuming their allocated drink will complete a 6 bouts of sprint interval exercise (10 second all-out maximal sprints interspersed with 50 seconds rest). Power output (peak and mean) during cycling sprints will be measured as the primary outcome measure. Salivary measures of nitrate/nitrite will be taken at three time points over the course of the morning on Day 5 - (i) pre-drink consumption; (ii) 2 hours post-drink consumption; and (iii) post-exercise. Plasma measures of nitrate and nitrite will be taken at two time points over the course of the morning on Day 5 - (i) pre-drink consumption; and (ii) 2 hours post-drink consumption. Near infra-red spectroscopy (NIRS) will be used to measure muscle (vastus lateralis) oxygenation during cycling bouts. A Stroop test to measure inhibition (executive function) will be taken pre- and post-exercise. Sensory perception of the drink will be measured immediately post-consumption on Day 5. After a 5-day washout period participants will crossover and begin their second trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21 - 40 years
* Healthy and injury-free (e.g., no cardiovascular disease, diabetes mellitus, orthopaedic impairment that interferes with moderate-to-vigorous exercise)
* Blood pressure < 130/90 mmHg
* Be physically active: Engaging in a minimum of 150 minutes of moderate-intensity exercise or 75 minutes of vigorous-intensity physical activity each week.
* Recreational cyclist (Minimum 1 hour cycling per week).
* Body mass index: 18.5-25 kg/m2
* Non-smoker
* Asian

Exclusion Criteria:

* Any allergies to beetroot or isotonic drink.
* Asthma
* Any diagnosed form of cardiometabolic disease (heart disease, stroke, peripheral vascular disease, diabetes, metabolic syndrome, high blood pressure).
* Any symptoms contraindicating exercise testing (e.g. chest pains).
* Any balance or dizziness problems.
* Any chronic medical conditions (whether medicated or not).
* Any bone joint problems.
* Any Physician diagnosed contraindications to exercise.
* Any other health problems that may be a cause for concern or contraindication to exercise.
* Any recent Covid vaccination (within last 2 weeks).

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Power output during maximal sprint cycling | 2 hours after drink ingestion
  Peak and mean power output

SECONDARY OUTCOMES:
Salivary nitrate | Pre-drink, 2 hours post-drink and immediately post-exercise (2.5 hours post-drink)
  Salivary nitrate/nitrite concentration
Plasma nitrate and nitrite | Pre-drink and 2 hours post-drink
  Plasma nitrate and nitrite
Muscle oxygenation | During exercise (2-2.5 hours post drink)
  Near infra-red spectroscopy
Sensory evaluation (Acceptance and Preference Test Evaluation by Meilgaard et al 2007) | Immediately post-drink (1 minute post-drink)
  Drink taste and perception (7-point scale - 1 extremely dislike to 7 extremely like)
Stroop test | Immediately pre- (2 hours post-drink) and immediately post-exercise (2.5 hours post drink)
  Reaction time and correct answers

CONTACTS AND LOCATIONS:
Locations (1):
- Human Bioenergetics Laboratory, National Institute of Education, Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
All published data will be placed into the Data Repository of Nanyang Technological University National Institute of Education for public access upon publication.
Supporting Information: Analytic Code
Time Frame: Upon publication - permanent repository
Access Criteria: Public repository - exact web address available upon publication.
URL: http://researchdata.nie.edu.sg/